CLINICAL TRIAL: NCT04044235
Title: HIV Incidence in a Cohort of and Evaluation of Pre-Exposure Prophylaxis for High Risk Adolescent Girls and Young Women in Urban Lilongwe, Central Malawi
Brief Title: Evaluation of Pre-Exposure Prophylaxis for High Risk Adolescent Girls and Young Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lighthouse Trust (Other)
Collaborators: United States President's Emergency Plan for AIDS Relief (U.S. Federal Agency); Ministry of Health, Malawi (Other Government); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Sam Phiri, PhD, MSc, DCM, Executive Director, Lighthouse Trust
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PrEP
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: A non- randomized study design being implemented in 2 facilities in Lilongwe Urban. The first component is a cross-sectional study of AGYW in which HIV testing counselors will offer HIV tests and assess HIV risk. A sample of AGYW testing HIV-negative and established to be at high risk will be consented to enroll in the PrEP study. In the second component, AGYW who refuse PrEP will be consented to enroll in an HIV incidence cohort study and will be followed every 3 months for 12 months to determine HIV incidence. In the third component, AGYW who consent will be enrolled in a PrEP study. The PrEP study has two phases, which are, (i) a formative qualitative study involving AGYW and PrEP providers to understand factors and barriers to delivering PrEP to AGYW and (ii) a feasibility study of delivering PrEP to HIV negative AGYW. AGYW will be followed every 3 months for 12 months to determine incidence, assess factors and costs of delivering PrEP to AGYW.
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PrEP Cohort (Experimental): AGYW HIV-negative and established to be at high risk will be consented to enroll in the PrEP study. AGYW will be followed every 3 months for 12 months to determine incidence, assess factors and costs of delivering PrEP to AGYW.
  Interventions: Behavioral: PrEP Cohort
- HIV Incidence (No Intervention): HIV Incidence Cohort: In the second component, AGYW who refuse PrEP will be consented to enroll in an HIV incidence cohort study and will be followed every 3 months for 12 months to determine HIV incidence.

INTERVENTIONS:
Behavioral: PrEP Cohort — AGYW who are eligible for PrEP will be educated about the risk and benefits. For AGYW (aged 18-24 years) who consent to PrEP, an ART provider (nurse or clinician) certified by the MOH will provide PrEP (package of disoproxil fumarate/emtricitabine (Truvada)) on the same day that the client is determined eligible. Peer navigators will ensure linkage to facilities for follow-up care. The initial follow-up visit will occur one month from PrEP initiation to ensure that the client is tolerating the regimen and to answer any questions, with three-month follow-up visits thereafter.
  Arms: PrEP Cohort

SUMMARY:
To provide preliminary evidence about feasibility and acceptability of delivering PrEP to AGYW identified as potentially at high risk of HIV infection in Lilongwe city communities and two public facilities in Lilongwe, Malawi. The primary objective of the study is to assess the feasibility, acceptability, tolerability and cost of delivering PrEP among high-risk AGYW aged 18-24 years and healthcare providers in urban Lilongwe. Secondary objectives are (i) to assess the program's ability to enroll and retain a PrEP cohort for one year and (ii) measure the incidence of HIV infection among high risk AGYW in urban Lilongwe among women who decline to enroll in the PrEP study (these will be offered enrollment in the HIV incidence study).

DETAILED DESCRIPTION:
The main goal of the study is to provide preliminary evidence about feasibility and acceptability of delivering PrEP to AGYW identified as potentially at high risk of HIV infection in Lilongwe city communities and two public facilities in Lilongwe, Malawi. The primary objectives are to; determine HIV prevalence among all AGYW identified as potentially at high risk of HIV infection in urban Lilongwe; assess the HIV program's ability to enroll and retain the PrEP cohort for one year; assess participants' and providers' perceptions of the barriers and facilitators for providing PrEP to inform implementation of PrEP study and future interventions and assess the cost of PrEP delivery in the routine HIV program.

Secondary Objectives:

1. To measure annual HIV incidence in a prospective cohort of HIV-negative AGYW identified as potentially at high risk of HIV infection but declined to enroll in PrEP cohort study in urban Lilongwe.
2. To measure annual HIV incidence among HIV-negative AGYW who enrolled in PrEP cohort study in urban Lilongwe.
3. To determine risk factors for HIV in a cohort of AGYW recruited in the prospective cohort study

ELIGIBILITY:
Inclusion Criteria:

Eligibility criteria for the cross-sectional study

* Female
* Consent to be counselled and tested for HIV
* Between 18 and 24 years old
* Ongoing HIV risk according to the risk Assessment guide
* Participated in the cross-sectional screening study or meets the eligibility criteria for the cross-sectional study
* Willing to provide written informed consent to participate in the HIV incidence study
* Accesses services at a mobile or fixed clinic in the defined catchment area
* Not planning to relocate in the next 12 months Eligibility criteria for the prospective PrEP for AGYW
* Participated in the cross-sectional study
* HIV-negative
* Answers yes to any two questions from the PrEP screening tool
* Willing and able to adhere to daily PrEP
* Willing to provide written informed consent to participate in the PrEP study
* Accesses services at a mobile or fixed clinic in the defined catchment area
* Not planning to relocate in the next 12 months

Eligibility criteria for focus group discussions for PrEP providers

* Provided PrEP for at least 3 months
* Trained nurse
* Orientated in PrEP and study procedures

Exclusion Criteria:

Exclusion criteria for the prospective HIV incidence phase

• HIV positive

Exclusion criteria for PrEP for AGYW

* Under 18 years or older than 24 years at enrollment (including AGYW aged 24 years at enrolment)
* Breastfeeding women
* Already taking oral or injectable PrEP through another study
* Current or past history of renal or liver disease
* Clients on multi-drug resistant tuberculosis (MDR-TB) medications
* Signs of acute HIV infection. The client would be asked to return after 3 months for a re-evaluation
* FSW <35kg
* Known allergy to tenofovir disoproxil fumarate (TDF) and/or emtricitabine (FTC);
* Unwilling or unable to return for 3-monthly HIV testing, counselling and safety monitoring visits or planning to relocate to another geographic area during the period of the study.
* Blood creatinine clearance (Cr Cl) <60ml/min

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1032 (Estimated)
Dates: Start 2019-06-25 (Actual); Primary Completion 2020-12-24 (Estimated); Study Completion 2020-12-24 (Estimated)

PRIMARY OUTCOMES:
Retention | 12 Months
  Proportion of participants by risk group and age enrollment who are retained at 3, 6, 9, 12 months after enrollment in each study arm
HIV Incidence | 12 Months
  Proportion of participants newly diagnosed HIV positive at 3, 6, 9, 12 months after enrollment in each study arm

SECONDARY OUTCOMES:
Follow-up outcomes | 12 months
  Number of participants by follow-up outcomes ( Discontinue, dead, withdraw, lost to follow-up) for each study arm
Uptake | 12 months
  Number of clients enrolled in each study arm

CONTACTS AND LOCATIONS:
Overall Officials: Sam Phiri, PhD, Principal Investigator — Lighthouse Trust
Locations (2):
- Malawi (2):
  - Bwaila Hospital, Lilongwe, Central Region
  - Kawale Health Centre, Lilongwe, Central Region

IPD SHARING:
Plan to Share IPD: No